CLINICAL TRIAL: NCT00377286
Title: Development of Biomarker and Functional Assessment Tools to Evaluate the Effect of Glucosamine on Joint Structure and Quality of Life
Brief Title: Effect of Glucosamine on Joint Structure and Quality of Life (JOG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: John Jakicic, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0604099
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee Pain; Glucosamine; MRI; CTX-II; Biomarkers; Skin quality
MeSH Terms: conditions — Osteoarthritis | interventions — Glucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): 1500 mg of lite lemonade
  Interventions: Other: 16 oz lite lemonade
- 1 (Active Comparator): 1500 mg glucosamine in 16 oz lite lemonade 1 time daily for 6 months
  Interventions: Dietary Supplement: Glucosamine (a dietary supplement)

INTERVENTIONS:
Dietary Supplement: Glucosamine (a dietary supplement) — 1500 mg in 16 oz lite lemonade, once per day for 6 months
  Arms: 1
Other: 16 oz lite lemonade — 16 oz lite lemonade 1 time daily for 6 months
  Other Names: Minute Maid
  Arms: 2

SUMMARY:
The goal of this study is 1) to develop a biomarker of of cartilage synthesis by determining if there is a relationship between changes in the status of knee cartilage and the amount of a biomarker called CTX-II in urine. 2) We will also characterize people who have experienced cartilage loss and/or reduced functional ability using performance tests and a questionnaire. 3) The administration of glucosamine in a beverage for six months will be used to promote the alteration in cartilage status and improve function in people with mild to moderate joint pain. A secondary goal will be to assess the effect of glucosamine on the skin in a small subset of women.

DETAILED DESCRIPTION:
Reduced knee function is a significant cause of physical limitations and disability. As cartilage deteriorates due to aging, wear-and-tear, injury, or disease, joint space narrowing and pain can develop. The lost of articular cartilage arises from an imbalance between cartilage synthesis and cartilage degradation. When cartilage needs to be remodeled, enzymes such as matrix metalloproteinases (MMPs) degrade type II collagen. It now may be possible to use new molecular markers of cartilage degradation to assess the progression of joint loss in comparison with radiographic changes of the knee joint. Urinary excretion of C-terminal cross linking telopeptide of type II collagen (CTX-II) is a new molecular marker of cartilage tissue degradation metabolism.

Recent evidence suggests that glucosamine, a dietary supplement, may provide some relief from joint pain and may increase the functional ability to participate in activities of daily living. This may be a result of these dietary supplements stimulating tissue repair such as cartilage in the affected joints, or by inhibiting the degradation of cartilage through an inhibition of enzymes. Moreover, Braham, Dawson, & Goodman (2003) reported increases in function in adults with knee pain following 12 -weeks of glucosamine supplementation. It is unclear, however, if glucosamine delivered via a liquid carrier would improve physical function and impact quality of life measures in people who have experienced loss of knee cartilage.

Glucosamine is a precursor for glycosaminoglycans, which are a major component of both joint cartilage and skin. Potential benefits of glucosamine on skin have been reported previously. It is possible that glucosamine in a beverage might also improve skin parameters over time.

Comparisons: 100 men and women with mild to moderate joint pain taking a liquid with glucosamine, compared to 100 men and women with mild to moderate joint pain taking a liquid with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female or male (female only for skin sub-study)
* 35-65 years of age (40 -65 for skin sub-study)
* Willingness to provide informed consent
* Willingness to be randomized to glucosamine or placebo
* Knee pain on more days than not for at least one month in past year
* Sum of WOMAC pain subscales between 300 and 500 inclusive
* Ability to read and understand English
* Ability to understand study procedures
* Dry skin for sub-study

Exclusion Criteria:

* Plans for elective surgery in the next 12 months Plans to move out of the area in the next 12 months
* Concurrent medical/arthritic disease that could confound or interfere with evaluation of pain or efficacy including inflammatory arthritis
* Spine or hip pain of sufficient magnitude to interfere with the evaluation of the knee
* Isolated patellofemoral disease manifested by primarily anterior knee pain in the absence of tibiofemoral radiographic finding
* History of arthroscopy of the affected knee within 6 months prior to study entry
* Allergy to,or history of significant clinical or laboratory adverse experience associated with acetaminophen or glucosamine
* Inability to undergo a MRI of knee
* Inability to walk without a cane or other assistive device
* Liver or kidney disease
* Diabetes mellitus
* Women who are currently pregnant or nursing, pregnant within the previous six months, or planning on becoming pregnant within the next 6 months
* Unwilling to use double barrier method of contraception
* Alcohol use in excess of 3 mixed drinks/day
* Corticosteroid treatment
* Sustained use of NSAIDS including aspirin in anti-inflammatory doses may be used for treatment of pain other than knee pain, if such use is intermittent
* Topical analgesics
* Other medical therapy for arthritis within one month prior to entry
* Participation in another clinical study with an investigational agent within the last 4 weeks
* Have taken glucosamine in past 3 months, chondroitin, Sam-E, MSM or other dietary supplements for knee pain within the past 6 months
* Have taken a bisphosphonate medication that affects bone turnover in the past 6 months
* Initiation of physical therapy or muscle conditioning program within 2 months prior to study entry
* Intra-articular injection of hyaluronic acid or congeners into the knee within past 12 months.
* Concurrent use of tetracycline, anticoagulants, dietary supplements or other complementary or alternative regimens for joint pain
* History of knee or hip replacement
* Weight exceeds 285 in men or 250 in women.
* Have had any of the following cancers: Acute Leukemia, Brain, Chronic Leukemia, Esophagus, Liver,Lung, Lymphoma, Multiple Myeloma, Pancreas, Skin Melanoma, and Stomach.
* Have taken any of the following doctor prescribed medications for arthritis: Methotrexate, Plaquenil, Hydroxychloroquine, Enbrel, Etanercept, Remicade, Infliximab, Arava, Leflunomide, Gold shots or pills, Prednisone pills, steroid pills, or glucocorticoid pills taken by mouth, Sulfasalazine, Kineret, Anakinra, Humira, and Adalimumab.
* Kellgren-Lawrence score of 4 (severe) in both knees based on x-ray.
* Anterior knee pain only with normal x-ray results.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of CTX-II at 3 and 6 months post intervention | 3 and 6 months
Measurement of bone marrow lesions, cartilage volume, as shown by MRI post intervention | 6 month

SECONDARY OUTCOMES:
Scores on WOMAC and KOOS of knee pain and function | 3 and 6 months
Scores on performance measures | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Jakicic, PhD, Principal Investigator — University of Pittsburgh; C. Kent Kwoh, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kwoh CK, Roemer FW, Hannon MJ, Moore CE, Jakicic JM, Guermazi A, Green SM, Evans RW, Boudreau R. Effect of oral glucosamine on joint structure in individuals with chronic knee pain: a randomized, placebo-controlled clinical trial. Arthritis Rheumatol. 2014 Apr;66(4):930-9. doi: 10.1002/art.38314. PMID 24616448
- [Derived] Roemer FW, Kwoh CK, Hannon MJ, Green SM, Jakicic JM, Boudreau R, Crema MD, Moore CE, Guermazi A. Risk factors for magnetic resonance imaging-detected patellofemoral and tibiofemoral cartilage loss during a six-month period: the joints on glucosamine study. Arthritis Rheum. 2012 Jun;64(6):1888-98. doi: 10.1002/art.34353. Epub 2011 Dec 27. PMID 22213129